CLINICAL TRIAL: NCT02884687
Title: Impact of Antimicrobial Stewardship in Hospital: Eight Years Review
Brief Title: Impact of Antimicrobial Stewardship in Hospital: Eight Years Review (BONANTIBIO)
Acronym: BONANTIBIO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-07Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Good Use of Antibiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study focuses on the use of antibiotics in Regional Hospital Center Metz-Thionville (CHRMT) between 2007 and 2014. To analyze the strategies and decisions related to the appropriate use of antibiotics for this center, some Semi-Directive Interviews (SDI) are realized on the study period with all concerned actors of the Good Use of antibiotics. An interviewing plan and tree interview guidelines were created. All SDI are processed by the same person.

DETAILED DESCRIPTION:
The study focuses on the use of antibiotics in Regional Hospital Center Metz-Thionville (CHRMT) between 2007 and 2014. CHRMT is a 2000-bed hospital in which 160 000 short hospitalizations are performed. To analyze the strategies and decisions related to the appropriate use of antibiotics for this center, some Semi-Directive Interviews (SDI) are realized on the study period with all concerned actors of the Good Use of antibiotics. An interviewing plan and tree interview guidelines were created. All SDI are processed by the same person.

ELIGIBILITY:
Inclusion Criteria:

* indication of antibiotics

Exclusion Criteria:

* Non Applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All antibiotics delivery
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evolution of the antibiotics use in the hospital compared with the efficacy indicators | 2007 to 2014

SECONDARY OUTCOMES:
Antibiotics consumption | 2007 to 2014
Bacterial resistance | 2007 to 2014
Composite index of the appropriate use of the antibiotics | 2007 to 2014

CONTACTS AND LOCATIONS:
Overall Officials: Gregory RONDELOT, MD, Study Director — CHR Metz-Thionville